CLINICAL TRIAL: NCT06768177
Title: Platelet Rich Plasma (PRP) as Terapeutical Option in Erectil Disfunction (DE)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: PRP vs CAVERJECT - 2023
Record Dates: First submitted 2024-12-03; First posted 2025-01-10 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Erectile Dysfunction Due to General Medical Condition; Erectile Dysfunction Following Radical Prostatectomy; Erectile Dysfunction Associated With Type 2 Diabetes Mellitus; Erectile Dysfunctions
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TREATMENT ARM (Experimental): 3 ML OF PRP
  Interventions: Drug: PRP injection
- COMPARISON ARM (Placebo Comparator): CAVERJECT 1 ML
  Interventions: Drug: Alprostadil 20 micrograms

INTERVENTIONS:
Drug: PRP injection — 3 ML OF PRP
  Arms: TREATMENT ARM
Drug: Alprostadil 20 micrograms — 1 ML
  Arms: COMPARISON ARM

SUMMARY:
Patients are randomized into 2 groups (A and B), subsequently group A is subjected to a cycle of 6 weekly injections of 3 ml of autologous PRP while group B is subjected to 6 weekly injections of 1 ml of caverject (alprostadil) 20 mcg. After 4 (four) weeks the groups will be crossed, so group A will be subjected to 6 weekly injections of 1 ml of caverject (alprostadil) 20 mcg while group B will be subjected to a cycle of 6 weekly injections of 3 ml of autologous PRP.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe erectile dysfunction (IIEF-5 score below 17)
* Patients previously treated with first- and second-line therapies for ED
* Patients who have undergone radical pelvic surgery with nerve sparing
* Good pharmacological blood pressure control
* Well-controlled diabetes on medication
* Current or former smokers
* Good renal function even with the use of medications
* Well-controlled hypertriglyceridemia and/or hypercholesterolemia even with the use of medications
* BMI less than or equal to 35
* Normal levels of FSH, LH, PRL, Total Testosterone, and TSH

Exclusion Criteria:

* Patients on antidepressant, anxiolytic, sedative, or antipsychotic medications.
* Consumers of more than 500 g of alcohol per day.
* BMI greater than 35
* Altered levels of FSH, LH, PRL, Total Testosterone, and TSH.

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in erectile function | 24 WEEKS
  Change in erectile function defined as the % of patients in each group achieving MCID in the IIEF-EF domain from baseline to 24 weeks (i.e. 12 weeks after the end of full treatment):
  * MCID (Minimal clinically important differences) is based on the severity of ED at baseline as:
  * Improvement of 5 or points more in IIEF score for patients with moderate ED (8-11) at baseline
  * Improvement of 2 or more points in IIEF score for patients with severe ED (5-7) at baseline

SECONDARY OUTCOMES:
EHS | 24 WEEKS
  Time frame: change from baseline and at 8 weeks, 16 weeks, and 24 weeks Any value above 0 (0 = The penis does not enlarge)
The percentage of patients in each group who achieve MCID in the IIEF-EF domain from baseline after treatment with PRP | 24 WEEKS
  MCID (Minimal Clinically Important Differences) is defined on the severity of ED at baseline as:
  * An improvement of 5 or more points in the IIEF score for patients with moderate ED (8-11) at baseline
  * An improvement of 2 or more points in the IIEF score for patients with severe ED (5-7) at baseline
The percentage of patients in each group who achieve MCID in the IIEF-EF domain from baseline after treatment with prostaglandin | 24 WEEKS
  MCID (Minimal Clinically Important Differences) is defined on the severity of ED at baseline as:
  * An improvement of 5 or more points in the IIEF score for patients with moderate ED (8-11) at baseline
  * An improvement of 2 or more points
The difference in the IIEF score from baseline to the end of treatment between the PRP group and the prostaglandin-treated group. | 24 WEEKS
  The difference in the IIEF score from baseline to the end of treatment between the PRP group and the prostaglandin-treated group.
SEP | 24 WEEKS
  Change in SEP:
  * Response to questions 2 and 3 (SEP-Q2: Were you able to insert your penis into your partner's vagina? / SEP-Q3: Did your erection last long enough to allow you to have successful intercourse?)
  * Change from baseline (= "YES" response) o At T1 (2 weeks after the end of the first cycle), T2 (2 weeks after the end of the second cycle), and T3 (3 months after the end of the complete treatment)
GAQ | 24 WEEKS
  Response to GAQ questions 1 and 2 (GAQ-Q1: Has the treatment you are taking improved your erectile function? / GAQ-Q2: If yes, has the treatment improved your ability to engage in sexual activity?) Change at T1 (2 weeks after the end of the first cycle), T2 (2 weeks after the end of the second cycle), and T3 (3 months after the end of the complete treatment) o Change from baseline (= "YES" response)
QEQ | 24 WEEKS
  At T1 (2 weeks after the end of the first cycle), T2 (2 weeks after the end of the second cycle), and T3 (3 months after the end of the complete treatment) o Improvement of 2 or more in the score
Change in EDITS between PRP vs. prostaglandins | At T1 (2 weeks after the end of the first cycle) and T2 (2 weeks after the end of the second cycle)
  At T1 (2 weeks after the end of the first cycle) and T2 (2 weeks after the end of the second cycle)
Change in TSS between PRP vs. prostaglandins | 3 months after the end of the complete treatment
  Change in TSS between PRP vs. prostaglandins at T3 (3 months after the end of the complete treatment)
Change in SHIM | 24 WEEKS
  Change in SHIM
  * At T1 (2 weeks after the end of the first cycle), T2 (2 weeks after the end of the second cycle), and T3 (3 months after the end of the complete treatment)
  * Improvement of 2 or more points in the score
ECDPD - Peak Systolic Velocity (PSV) | 24 WEEKS
  ECDPD - Peak Systolic Velocity (PSV):
  * To assess penile hemodynamics from baseline to T1 (2 weeks after the end of the first cycle), T2 (2 weeks after the end of the second cycle), and T3 (3 months after the end of the complete treatment)
  * Recording of arterial penile velocity (cm/s) o Improvement in cm/s (any > 30 cm/s)
ECDPD - Resistance Index (RI) | 24 WEEKS
  ECDPD - Resistance Index (RI):
  * To assess penile hemodynamics from baseline to T1 (2 weeks after the end of the first cycle), T2 (2 weeks after the end of the second cycle), and T3 (3 months after the end of the complete treatment)
  * Penile vascular resistance index (ratio) o Improvement (any increase up to the normal value - 0.9)
ECDPD - End-Diastolic Velocity (EDV) | 24 WEEKS
  ECDPD - End-Diastolic Velocity (EDV):
  * To assess penile hemodynamics from baseline to T1 (2 weeks after the end of the first cycle), T2 (2 weeks after the end of the second cycle), and T3 (3 months after the end of the complete treatment)
  * Recording of residual flow in a vessel at the end of the diastolic phase (cm/s)
  * Improvement in cm/s (any decrease in cm/s)
Adverse events | 24 WEEKS
  Adverse events: Number of participants who experienced treatment-related adverse events.
  Defined as: skin reaction (e.g., swelling, erythema, and warmth), discomfort at the injection site, penile pain, change in penile appearance, new sexual problems, and any systemic reaction observed by investigators or concerns expressed by patients o At T1 (2 weeks after the end of the first cycle), T2 (2 weeks after the end of the second cycle), and T3 (3 months after the end of the complete treatment)

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico di Bari - Azienda Ospedaliero Universitaria Consorziale Policlinico, Bari, Italy

IPD SHARING:
Plan to Share IPD: Undecided